CLINICAL TRIAL: NCT02468284
Title: An Open-label, Multi-Centre Trial Investigating Pharmacokinetics of Degarelix After a Starting Dose of 240 mg (40 mg/mL) Followed by Six Maintenance Doses of 80 mg (20 mg/mL) in Chinese Patients With Prostate Cancer Requiring Androgen Deprivation Therapy
Brief Title: Pharmacokinetics of Degarelix in Chinese Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 000200
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental)
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix
  Other Names: Firmagon

SUMMARY:
The purpose of this trial is to look at how much a new trial drug get into body, such as when the drug concentration in your body reaches peak and how high the peak value is.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed (Gleason graded) adenocarcinoma of the prostate (all stages), for which endocrine therapy (except for neoadjuvant hormonal therapy) is indicated
* Has a Prostate-specific Antigen (PSA) level ≥2.0 ng/mL at Screening
* Has a screening serum testosterone level >150 ng/dL
* Has an Eastern Cooperative Oncology Group (ECOG) score of ≤2

Exclusion Criteria:

* Has had previous or is currently under hormonal management of prostate cancer. However, hormonal therapy for a maximum duration of 6 months is accepted. This treatment should have been terminated at least 6 months prior to the Screening Visit
* Is currently treated with a 5-alpha reductase inhibitor
* Is considered to be candidate for curative therapy, i.e. radical prostatectomy or radiotherapy
* Is in need of neoadjuvant hormonal therapy
* Has a history of bilateral orchiectomy, adrenalectomy, or hypophysectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration observed (Cmax) | Day 0 - 196
Time of Cmax after subcutaneous administration (Tmax) | Day 0 - 196
Maximum plasma concentration observed (Cmax) | Day 0 - 28
Maximum plasma concentration observed (Cmax) | Day 168 - 196
Time of Cmax after subcutaneous administration (Tmax) | Day 0 - 28
Time of Cmax after subcutaneous administration (Tmax) | Day 168 - 196
Area under the plasma concentration-time curve during a drug dosing interval (AUC) | Day 0 - 28
Area under the plasma concentration-time curve during a drug dosing interval (AUC) | Day 168 - 196

SECONDARY OUTCOMES:
Plasma trough levels of degarelix | At Days 28, 56, 168 and 196

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Peking University Third Hospital (there may be other sites in this country), Beijing, China